CLINICAL TRIAL: NCT06429605
Title: Evaluating the Efficacy and Safety of Preoperative Administration of Duloxetine for Pain Management in Women Undergoing Hysterectomy Via Vaginal Route
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, MD., Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Muğla-77
Record Dates: First submitted 2024-05-15; First posted 2024-05-28 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Vaginal Hysterectomy; Postoperative Pain; vNOTES
MeSH Terms: conditions — Pain, Postoperative | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Only our clinic's standard preoperative and postoperative care were used (Güngördük K, Selimoğlu B, Gülseren V, Yasar E, Comba C, Özdemir İA. Effect of abdominal hot pack application on gastrointestinal motility recovery after comprehensive gynecologic staging surgery. Int J Gynaecol Obstet. 2024 Mar;164(3):1108-1116)
- Duloxetine (Experimental): In addition to our standard clinical protocol, study patients were administered 60 mg oral duloxetine 2 hours before surgery and 24 hours after surgery
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — In addition to our standard clinical protocol, study patients were administered 60 mg oral duloxetine 2 hours before surgery and 24 hours after surgery
  Arms: Duloxetine

SUMMARY:
Hysterectomy performed through the vaginal route (HVR) is the preferred method for women seeking hysterectomy to address uterine concerns such as premalignant conditions and fibroids. Compared to abdominal or laparoscopic approaches, HVR has shown to lead to quicker recovery times and faster resumption of daily activities. However, effectively managing postoperative pain remains a significant challenge for HVR patients.

Duloxetine, a serotonin-norepinephrine reuptake inhibitor typically prescribed for major depression and anxiety, has also been utilized in treating chronic pain conditions like osteoarthritis and musculoskeletal pain. However, research into its use for alleviating acute postoperative pain is currently limited to a single trial. Additionally, it's unclear whether perioperative duloxetine could enhance overall recovery quality after surgery. This study hypothesized that perioperative duloxetine could improve postoperative recovery for HVR patients, with evaluation using the Quality of Recovery-15 questionnaire (QoR-15).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing HVR ( vaginal natural orifice transluminal endoscopic surgery) hysterectomy and salpingectomy, with the option of additional procedures such as oophorectomy, uterosacral ligament plications, trans obturator tape insertion, colporrhaphy, or sentinel lymphadenectomy
* American Society of Anesthesiologists grade 1-3

Exclusion Criteria:

* patients with chronic non-gynecologic conditions (liver-renal or pulmonary disease)
* those using psychiatric drugs (antidepressants, neuroleptics, lithium) in the last 1 year,
* those with duloxetine allergy
* those using opioids for gynecologic or non-gynecologic conditions
* additional concurrent abdominal procedures
* Total vaginal prolapsus (POPQ 4)

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
The primary outcome | 8 hours after surgery
  the level of abdominal pain during ambulation (according to VAS score) Since the visual analog scale (VAS) has been used in prior studies for evaluating similar outcomes [10], a 100-mm VAS was used to grade the level of pain. For assessing pain at rest, patients were asked to grade their level of pain from 0 (no pain) to 10 (worst pain ever experienced) at the abdomen and at the vagina while lying in bed. For assessing pain during ambulation, patients were asked to stand up, walk a few steps, and sit in a chair. Then, they were asked to grade their pain, using the same scale, during ambulation.

SECONDARY OUTCOMES:
total QoR-15 score. | on postoperative day 2
  The QoR-15 is a 15-item questionnaire that measures the patient's QoR. Each item is answered on an 11-point numerical rating scale. The score ranges from 0 to 150 with a higher score indicating a better QoR. It measures in the domains of pain, physical comfort, physical independence, psychological support, and emotional state

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Education and Research Hospital, Muğla, Turkey (Türkiye)